CLINICAL TRIAL: NCT03299894
Title: Usefulness of Routine qSOFA Calculation at Triage to Fasten Antimicrobial Administration in Patients With Bacterial Infection in the Emergency Department: a Quasi-experimental Study
Brief Title: Impact of qSOFA Calculation on the Timing of Antimicrobial Therapy in the Emergency Department
Acronym: qSOFAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRO 2017-06
Record Dates: First submitted 2017-09-25; First posted 2017-10-03 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Bacterial Infection; Intensive Care
Keywords: Sepsis; Shock, septic; Emergency service, hospital; Anti-infective agents; Outcome assessment
MeSH Terms: conditions — Bacterial Infections; Sepsis; Shock, Septic; Emergencies

STUDY DESIGN:
Intervention Model Description: Patients will be prospectively included at Emergency Department triage during 2 consecutive 6-month periods (1-month wash-out interlude between the 2 inclusion periods):
  * First inclusion period: usual procedures for patient triage at Emergency Department admission and management of suspected or proven bacterial infection.
  * Second inclusion period: usual procedure for patient triage at Emergency Department admission PLUS routine calculation of qSOFA in all patients admitted to the Emergency Department with a suspected or proven bacterial infection. Patients with a qSOFA value ≥2 will be directly and immediately notified to Emergency Department physicians by triage nurses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- systematic calculation of qSOFA (Experimental): Usual procedure for patient triage AND systematic calculation of qSOFA at Emergency Department triage in patients admitted with a suspected or proven bacterial infection.
  Interventions: Procedure: systematic calculation of qSOFA
- no systematic calculation of qSOFA (No Intervention): Usual procedures for patient triage at Emergency Department admission and management of suspected or proven bacterial infection. No systematic calculation of qSOFA.

INTERVENTIONS:
Procedure: systematic calculation of qSOFA — calculation of qSOFA for each patient
  Arms: systematic calculation of qSOFA

SUMMARY:
The delayed administration of an adequate antimicrobial therapy is a strong predictor of impaired outcome in patients with bacterial sepsis. Therefore, the current Surviving Sepsis Campaign guidelines (2016) recommend that administration of intravenous antimicrobials be initiated within one hour following the recognition of sepsis or septic shock.

The quick Sepsis-related Organ Failure Assessment (qSOFA) score is a new bedside tool which has been recently proposed by the Third International Sepsis Consensus Definitions Task Force (Sepsis-3) to identify patients with suspected infection who are at greater risk for a poor outcome outside the Intensive Care Unit (ICU). It uses three criteria, assigning one point for low systolic blood pressure (SBP ≤100 mmHg), high respiratory rate (≥22 breaths per min) and altered mentation (Glasgow coma scale <15). The score ranges from 0 to 3 points. A qSOFA value ≥2 points is associated with a greater risk of death or prolonged ICU stay, these outcomes being more common in infected patients who may be septic than in those with uncomplicated infection. The definite goal of qSOFA is to hasten the management and thus improve the outcome of patients at risk of sepsis or septic shock.

Many patients admitted to the hospital for bacterial sepsis or septic shock are initially managed in the Emergency Department (ED). This study aims at investigating whether the routine calculation of qSOFA at patient triage may hasten the initiation of antimicrobial therapy in patients admitted to the ED with suspected or proven bacterial infection, especially in those with subsequent criteria for sepsis or septic shock (Sepsis-3 definition).

ELIGIBILITY:
Inclusion Criteria:

• Suspected or proven bacterial infection at emergency department triage

Exclusion Criteria:

* Imminent death
* Pregnancy
* Breast-feeding
* For patients managed by a medicalized pre-hospital emergency team before ED admission : administration of a first dose of antimicrobial agent before ED admission
* Lack of coverage by the public health insurance system
* Patient's refusal for study enrollment
* Lack of confirmed bacterial infection (i.e., documented either clinically, microbiologically or by imaging procedures) in patients with a suspected bacterial infection at emergency departement triage

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-06-10 (Actual); Study Completion 2018-06-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who receive a first dose of antimicrobial agent | one hour
  Proportion of patients with criteria for sepsis or septic shock (Sepsis-3 definition) who receive a first dose of antimicrobial agent within one hour following triage in the emergency department.

SECONDARY OUTCOMES:
Proportion of patients who receive a first dose of adequate antimicrobial agent | one hour
  Proportion of patients with criteria for sepsis or septic shock (Sepsis-3 definition) and microbiologically documented infection who receive a first dose of adequate antimicrobial agent within one hour following triage in the emergency department.
Proportion of patients who receive a first dose of antimicrobial agent | three hours
  Proportion of patients with criteria for sepsis or septic shock (Sepsis-3 definition) who receive a first dose of antimicrobial agent within 3 hours following triage in the emergency department.
Proportion of patients who receive a first dose of adequate antimicrobial agent | three hours
  Proportion of patients with criteria for sepsis or septic shock (Sepsis-3 definition) and a microbiologically documented infection who receive a first dose of adequate antimicrobial agent within 3 hours following triage in the emergency department
Proportion of patients with a decrease in SOFA score value ≥ 1 point | two days
  Proportion of patients with a decrease in SOFA score value ≥ 1 point between triage in the emergency department (Day 0) and Day 2 among those with an initial SOFA score value ≥ 1 point
Proportion of patients requiring an admission to the Intensive Care Unit | two days
  Proportion of patients requiring an admission to the Intensive Care Unit between triage in the emergency department (Day 0) and Day 2
In-hospital mortality at day 7 | seven days
  Number of patients who died in hospital at day 7
Overall In-hospital mortality | through hospital discharge, up to 3 months
  Number of patients who died in hospital during the hospital stay
Length of hospital stay | throught hospital discharge, up to 3 months
  Number of days in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Julien PASSERIEUX, MD, Principal Investigator — Regional Hospital Center of Orleans
Locations (1):
- Regional Hospital center of Orleans, Orléans, France

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Derived] Petit J, Passerieux J, Maitre O, Guerin C, Rozelle C, Cordeau O, Cassonnet A, Malet A, Boulain T, Barbier F; qSOFAST study group. Impact of a qSOFA-based triage procedure on antibiotic timing in ED patients with sepsis: A prospective interventional study. Am J Emerg Med. 2020 Mar;38(3):477-484. doi: 10.1016/j.ajem.2019.05.022. Epub 2019 May 10. PMID 31103379